CLINICAL TRIAL: NCT02668926
Title: Endocrine and Emotional Effects of Lisdexamfetamine and d- Amphetamine: a Placebo-controlled Study in Healthy Subjects (LisDexStudy)
Brief Title: Endocrine and Emotional Effects of Lisdexamfetamine and d-Amphetamine.
Acronym: LisDex
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: EKNZ 2015-00015
Record Dates: First submitted 2016-01-21; First posted 2016-01-29 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Healthy
MeSH Terms: interventions — Lisdexamfetamine Dimesylate; Dextroamphetamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Lisdexamfetamine, d-amphetamine, Placebo (Experimental): Cross-over within-subjects design with all treatment conditions tested in the same subject. This design has 3 arms with three treatment conditions in the same subject. The three treatment conditions are placebo, lisdexamfetamine, and d-Amphetamine sulfate.
  Interventions: Drug: Lisdexamfetamine, d-amphetamine, Placebo
- d-amphetamine, Placebo, Lisdexamfetamine (Experimental): Cross-over within-subjects design with all treatment conditions tested in the same subject. This design has 3 arms with three treatment conditions in the same subject. The three treatment conditions are placebo, lisdexamfetamine, and d-Amphetamine sulfate.
  Interventions: Drug: d-amphetamine, Placebo, Lisdexamfetamine
- Placebo, Lisdexamfetamine, d-amphetamine (Experimental): Cross-over within-subjects design with all treatment conditions tested in the same subject. This design has 3 arms with three treatment conditions in the same subject. The three treatment conditions are placebo, lisdexamfetamine, and d-Amphetamine sulfate.
  Interventions: Drug: Placebo, Lisdexamfetamine, d-amphetamine

INTERVENTIONS:
Drug: Lisdexamfetamine, d-amphetamine, Placebo — Elvanse (Lisdexamfetamine): 100mg p.o, single dose; d-Amphetamine: 40.3mg p.o, single dose; Placebo: Capsules containing mannitol looking identical to lisdexamphetamine and d-Amphetamine.
  Other Names: Lisdexamfetamine=Elvanse, d-amphetamine=d-amphetamine sulfate
  Arms: Lisdexamfetamine, d-amphetamine, Placebo
Drug: d-amphetamine, Placebo, Lisdexamfetamine — Elvanse (Lisdexamfetamine): 100mg p.o, single dose; d-Amphetamine: 40.3mg p.o, single dose; Placebo: Capsules containing mannitol looking identical to lisdexamphetamine and d-Amphetamine.
  Other Names: Lisdexamfetamine=Elvanse, d-amphetamine=d-amphetamine sulfate
  Arms: d-amphetamine, Placebo, Lisdexamfetamine
Drug: Placebo, Lisdexamfetamine, d-amphetamine — Elvanse (Lisdexamfetamine): 100mg p.o, single dose; d-Amphetamine: 40.3mg p.o, single dose; Placebo: Capsules containing mannitol looking identical to lisdexamphetamine and d-Amphetamine.
  Other Names: Lisdexamfetamine=Elvanse, d-amphetamine=d-amphetamine sulfate
  Arms: Placebo, Lisdexamfetamine, d-amphetamine

SUMMARY:
The study will compare the acute emotional and endocrine effects of equivalent doses of lisdexamfetamine and amphetamine in healthy subjects. In addition the pharmacokinetics and effects of the amphetamines on aspects of social cognition are investigated.

ELIGIBILITY:
Inclusion Criteria:

healthy subjects aged 18-45 years

Exclusion Criteria:

1. Chronic or acute medical condition including clinically relevant abnormality in physical exam, laboratory values, or ECG.
2. Current or previous psychotic or major affective disorder
3. Psychotic or major affective disorder in first-degree relatives
4. Prior illicit drug use (cannabis) more than 5 times or any time within the previous 2 months.
5. Pregnant or nursing women.
6. Participation in another clinical trial (currently or within the last 30 days)
7. Use of medications that are contraindicated or otherwise interfere with the effects of the study medications (monoamine oxidase inhibitors, antidepressants, sedatives etc.)
8. Tobacco smoking (>10 cigarettes/day)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-05; Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Effects of lisdexamphetamine and d-Amphetamine on circulating steroidal hormones | 13 hours
  Measurement of different circulating hormones before and after drug
Subjective effects of lisdexamphetamine and d-amphetamine | 13 hours
  Assessment of subjective effects using visual analog scales

SECONDARY OUTCOMES:
Effects of lisdexamphetamine and d-Amphetamine on emotion recognition and empathy | 1h
  Assessment of emotion recognition and empathy using different Computer Tasks.

OTHER OUTCOMES:
Pharmacokinetics | 13h
  Collection of blood samples for measurement of plasma concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Matthias E Liechti, MD, MAS, Principal Investigator — University Hospital, Basel, Switzerland; Alex Odermatt, Dr., Study Chair — University of Basel
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dolder PC, Strajhar P, Vizeli P, Odermatt A, Liechti ME. Acute effects of lisdexamfetamine and D-amphetamine on social cognition and cognitive performance in a placebo-controlled study in healthy subjects. Psychopharmacology (Berl). 2018 May;235(5):1389-1402. doi: 10.1007/s00213-018-4849-0. Epub 2018 Feb 9. PMID 29511807
- [Derived] Dolder PC, Strajhar P, Vizeli P, Hammann F, Odermatt A, Liechti ME. Pharmacokinetics and Pharmacodynamics of Lisdexamfetamine Compared with D-Amphetamine in Healthy Subjects. Front Pharmacol. 2017 Sep 7;8:617. doi: 10.3389/fphar.2017.00617. eCollection 2017. PMID 28936175